CLINICAL TRIAL: NCT05976529
Title: Efficacy and Safety of Dydrogesterone After Operation of Ovarian Endometrial Cysts: a Multicenter, Observational Clinical Study
Brief Title: A Multicenter, Observational Clinical Study of Dydrogesterone
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Women and Children Hospital (Other)
Responsible Party: Principal Investigator, Li Li, Deputy Director, Institute of Women's and Children's Health, Guangdong Women and Children Hospital
Other Study IDs: GuangdongWCH-LiLi02
Record Dates: First submitted 2023-04-25; First posted 2023-08-04 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Endometriosis; Endometriosis Ovary
Keywords: endometriosis; dydrogesterone; therapeutic effect evaluation; safety; dienogest
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: From the 5th to 25th day of menstrual cycle, 10 mg dydrogesterone was taken orally twice a day for 3 menstrual cycles.
- control group: After postoperative pathological diagnosis, oral dienogest was started, 4 weeks as a course of treatment, and 3 courses of continuous treatment were given.

SUMMARY:
The objective of this study was to investigate the efficacy and safety of dydrogesterone in the long-term management of ovarian endometriosis cyst after surgery.

DETAILED DESCRIPTION:
Endometriosis refers to the appearance, growth and infiltration of endometrial tissue (glands and stroma) in the lining of the uterine cavity and other parts of the uterus, and repeated bleeding, which causes pain, infertility and nodules or masses. Endometriosis is a common gynecological disease in Chinese female patients, and its incidence has been increasing in recent years, which seriously affects the fertility and quality of life of patients. The typical clinical manifestations of endometriosis mainly include dysmenorrhea, pelvic pain and dyspareunia. Dysmenorrhea is a common symptom of endometriosis, which is secondary and persistent. The pain is most severe on the first day of menstruation and disappears completely at the end of menstruation. Pain is mainly caused by endometriosis bleeding, which irritates the inflammatory response of local tissues. Endometriosis lesions secrete prostaglandins, which cause contracture of uterine muscles and aggravate dysmenorrhea. Ovarian endometriotic cysts are the most common and easily detected type of endometriosis. Its clinical manifestations include: 1) dysmenorrhea, affecting daily activities and life; 2) chronic pelvic pain; 3) pain during or after sexual intercourse; 4) often complicated with infertility; 5) ovarian endometriotic cyst formation by imaging examination; 6) elevated CA125.

According to the guidelines for the diagnosis and treatment of endometriosis (third edition) published by Chinese Journal of Obstetrics and Gynecology in December 2021, ovarian endometriosis cysts can be divided into medical treatment and surgical treatment. The indications for drug therapy were: 1) ovarian endometriosis cyst diameter <4cm; 2) have pelvic pain. The treatment drugs include oral contraceptives, progesterone analogues, gestrinone, gonadotropin-releasing hormone agonist (GnRHa) and traditional Chinese medicine. The indications for surgical treatment were: 1) the diameter of ovarian endometriosis cyst ≥4cm; 2) combined infertility; 3) pain medications are ineffective. In clinical practice, most patients lose the opportunity of drug treatment, or drug treatment is ineffective, and most patients need surgical treatment. Laparoscopic surgery is the first choice for surgical treatment, and cystectomy is recommended. However, surgical treatment can only remove the superficial lesions, and it is difficult to remove the deep lesions, which is easy to leave lesions. After surgery, affected by steroid hormones, the small lesions left are easy to relapse, leading to the characteristics of recurrent disease. Therefore, the recurrence rate of ovarian endometriosis cyst after conservative surgery is high, and it must be treated with drugs and long-term management after surgery.

In the postoperative drug management of ovarian endometriosis cyst, the first-line drugs are mainly progesterone analogues (dienogest), GnRH-a, dydrogesterone and so on. There is evidence that the continuous use of dienogest for 24 months after surgery can significantly reduce the recurrence rate of ovarian endometriosis cysts. Dienogest is a fourth-generation highly selective progesterone receptor agonist, which acts locally on endometriotic lesions, has no male, estrogen, glucose and mineralocorticoid activity, and does not affect metabolism. It is used in the first-line treatment of endometriosis. "In a German retrospective study, dienogest 2 mg daily for 60 months was effective in reducing endometriosis associated pelvic pain, and dienogest was well tolerated." However, ovulation was inhibited in most patients during dienogest treatment. For patients with fertility needs, menstruation returned to normal after stopping dienogest for 2 months. To pregnant element is the most common adverse drug reactions: frequent or long time of uterine bleeding (3.2%), insomnia (2.7%), acne (2.1%), nausea (2.1%), weight (2.1%), lower abdominal discomfort (1.6%), headache (1.6%), breast discomfort (1.1%), and depressed mood (1.1%). Therefore, it is not suitable to use dienogest for postoperative management in patients with ovarian endometriosis who are in urgent need of pregnancy after surgery. At present, the cost of dienogest in our country is relatively high, about 500 yuan for a box (28 tablets), and there will be a certain economic burden for ordinary patients.

"Dydrogesterone is similar in structure to conventional progesterone and has only progestogen activity without estrogen, androgen, or mineralocorticoid activity. It atrophies the ectopic endometrium, prevents the development of new endometriotic lesions, and does not inhibit normal endometrium or ovulation. The menstrual cycle is regular in the course of regular treatment with dydrogesterone, so normal pregnancy can be achieved during the treatment." An open, multi-center, post-marketing, observational clinical study in Japan showed that dydrogesterone could effectively inhibit the growth of ovarian endometriosis cysts and improve the total score of dysmenorrhea and the degree of dysmenorrhea pain. Studies have shown that long-term treatment of endometriosis with dydrogesterone after surgery for 12 months can significantly reduce endometriosis-associated pain, treat infertility, and prevent recurrence of the disease. A Japanese multi-center study showed that the incidence of adverse drug reactions of dydrogesterone was 31.8%, and the most common adverse event was uterine bleeding. Dydrogesterone endometriosis was effective, safe and clinically beneficial for patients. For patients in urgent need of pregnancy, natural pregnancy can still be achieved during postoperative medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had undergone laparoscopic ovarian cyst excision and were confirmed by pathological diagnosis as ovarian endometriosis cyst (pathology was completed in each central hospital).
* Ovarian cyst >4cm.
* Concomitant infertility.
* Patients who fail to respond to medication.
* American Society of Reproductive Medicine(ASRM) stages were II-IV.
* No relevant therapeutic drugs, such as dydrogesterone, dienogest, GnRHa, etc., were used 3 months before treatment.
* No combined endocrine diseases.

Exclusion Criteria:

* Ovulation disorders, immune defects and genital development abnormalities caused by infertility.
* Patients who are allergic to the drugs used in this study.
* Patients with severe hepatorenal insufficiency or malignant tumor.
* Those who took hormone medication within 3 months before the study date.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Patients aged 18-45 years after surgery for ovarian endometriosis cyst
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual analogue pain score(VAS) | before drug treatment and 3 months after drug treatment
  The visual analogue scale (VAS) was used to evaluate the pain. It is widely used in clinical practice in China. The basic method is to use a swimming ruler of about 10cm in length, marked with 10 scales on one side, and "0" and "10" points on both ends, with 0 points indicating no pain and 10 points indicating the most severe pain that can be endured.
Endometriosis fertility index(EFI) | before drug treatment and 3 months after drug treatment
  EFI score of endometriosis refers to the evaluation of fertility in patients with normal semen in men and good ovarian reserve function in women without adenomyosis. The pregnancy rate was measured by quantifying the patient's age, the duration and type of infertility, and the function of the fallopian tubes, uterus, and ovaries. If the score is higher than 9, the patient can try natural pregnancy. If the score is 5-8 points, the patient can be monitored by fertility guidance, if not naturally pregnant, can be treated by IVF-ET. If the score is lower than 5 points, the patients can be directly treated by IVF-ET.
The Cox Menstrual Symptom Scale(CMSS) | before drug treatment and 3 months after drug treatment
  The Cox menstrual symptom scale (CMSS) was used to evaluate the severity of symptoms and the duration of dysmenorrhea. The scale included 2 parts, CMSS-severity (CMSS-S) and CMSS-duration (CMSS-T), with a total of 18 observation indicators. It included 17 symptoms including nausea, vomiting, loss of appetite, headache, vertigo and the duration of dysmenorrhea. All CMSS-S items were scored on a 5-point scale: 0 as no symptoms, 1 as mild, 2 as moderate, 3 as severe, and 4 as extremely severe. CMSS-T is also a 5-point scale: 0 for no symptoms, 1 for persistent < 3h, 2 for 3~7h, 3 for 7~24h, 4 for continuous > 24 hours.

SECONDARY OUTCOMES:
Serum CA125 | before drug treatment and 3 months after drug treatment
  In some infectious diseases, autoimmune diseases, gynecological benign diseases, malignant tumors can appear CA125 significantly increased.
Anti-mullerian hormone(AMH) | before drug treatment and 3 months after drug treatment
  AMH is an important index to evaluate AMH is an important index to evaluate the reserve function of ovarian.
Short form 36（SF36） | before drug treatment and 3 months after drug treatment
  The SF36 is a short questionnaire with 36 items which measure eight multi-item variables: physical functioning (10 items), social functioning (two items), role limitations due to physical problems (four items), role limitations due to emotional problems (three items), mental health (five items), energy and vitality (four items), pain (two items), and general perception of health (five items). There is a further unscaled single item on changes in respondents' health over the past year. For each variable item scores are coded, summed, and transformed on to a scale from 0 (worst possible health state measured by the questionnaire) to 100 (best possible health state).
The postoperative pregnancy of the patients. | 3 months after drug treatment
  Patients were followed up by phone calls to find out whether they were pregnant.

OTHER OUTCOMES:
Liver function | before drug treatment and 3 months after drug treatment
  Liver function is used to assess the safety level of dydrogesterone and dienogest. Liver function includes the level of ALT, AST, ALT/AST by blood test.
Kidney function | before drug treatment and 3 months after drug treatment
  Kidney function is used to assess the safety level of dydrogesterone and dienogest. Kidney function includes the level of Urea, CO2, CRE, UA, β2-MG by blood test.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Yuan, Master, Principal Investigator — Guangdong Women and Children Hosptial
Locations (1):
- Guangdong Women and Children Hospital, Guanzhou, Guangdong, China